CLINICAL TRIAL: NCT04078399
Title: Efficacy and Safety of Azacitidine Combined With Interferon in the Treatment of Recurrence of Allogeneic Hematopoietic Stem Cell Transplantation in Myeloid Tumors of the Blood System
Brief Title: Efficacy and Safety of Azacitidine Combined With Interferon in the Treatment of Post-transplant Recurrence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY- aza-relapse-2019002
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: HSCT; Efficacy and Safety
Keywords: azacitidine; HSCT; interferon; safety; Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with recurrence after allogeneic transplantat (Experimental): One arm
  Interventions: Drug: Azacitidine combined with interferon preemptive treatment

INTERVENTIONS:
Drug: Azacitidine combined with interferon preemptive treatment — Azacitidine combined with interferon preemptive therapy for prevention and treatment of recurrence of allogeneic transplantation of myeloid tumors (AML/MDS/MPN) in the blood system

SUMMARY:
This study is a single-center, one-arm, prospective, phase II clinical trial with the primary objective of assessing the effectiveness of azacitidine combined with interferon in the prevention of recurrence after allogeneic transplantation of myeloid tumors (AML/MDS/MPN) in the blood system. Sex and safety.

At the screening/baseline period, informed consent is obtained and the inclusion/exclusion criteria are checked. Plan to enroll 30 patients, and collect demographic data, medical history data, vital signs, physical examination, laboratory tests (hematuria, liver and kidney function; immune indicators: T cell subsets, Treg, etc.), pregnancy test for female patients And other necessary auxiliary inspections.

The time to start treatment is: a decrease in chimerism and/or minimal residual disease (MRD) after myeloid tumor allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Treatment programs:

1. Basic protocol: Azacitidine is administered subcutaneously at 32 mg/m2/d for 5 consecutive days; α-interferon treatment started on day 8 for 3 weeks; 4-6 weeks/treatment with long-acting interferon Gebin). 1-1.5 million U / kg, once a week; or ordinary alpha-interferon, 200 acres / square meter / d (total ≥ 300MU / d), 5-7 days a week;
2. Start time of medication:

1 In the absence of immunosuppressive agents such as cyclosporine, the chimeric rate is decreased and/or MRD-positive: or in the case of immunosuppressive agents such as cyclosporine, the chimeric rate is fully chimeric and MRD-positive: A-interferon is first administered. Single-agent intervention, if there was no significant decrease in MRD for 2 consecutive courses (MRD decreased ≤ 50%), azacitidine combined with interferon intervention was started; 2 In the case of calmodulin immunosuppressant (cyclosporine or tacrolimus), the chimeric rate decreased and the MRD was negative, the immunosuppressant was rapidly reduced or discontinued, and the bone marrow was reviewed 2 weeks, if the chimeric rate did not rise. (decreased or stable), or after two consecutive immunosuppressive adjustments did not reach complete chimerism, start azacitidine combined with interferon intervention; (3) If cyclosporine or other immunosuppressive agents are applied before the start of the study, rapid reduction; dose reduction 1 / 4-1 / 2; if the chimeric rate increases or GVHD occurs, continue the immunosuppressant adjustment strategy; (4) Stop treatment: acute GVHD above II degree; patients are intolerant to the study protocol; basic regimen is ineffective after 2 courses of treatment (chimeric rate continues to decline or MRD continues to increase) or disease recurrence; transplant.

ELIGIBILITY:
Inclusion criteria:

Patients enrolled must meet the following criteria:

1. ≥ 14 years old, male or female;
2. Patients with allogeneic peripheral blood stem cell transplantation due to myeloid tumors of the blood system (AML/MDS/CML/MPN, etc.);
3. Recurrence trend evaluation criteria: the proportion of bone marrow blast cells <5%; flow cell MRD ≥ 0.01% and interval 2 consecutive times 2 times; fusion gene interval 2 weeks at least 2 consecutive positive and rising trend or from negative to positive; Bone marrow WT1 levels increased dynamically and were greater than 0.6%; chimeric rate (STR) decreased by >5% (STR <90%) or XY-FISH donor chimerism decreased by >0.5%;
4. Blood routine: neutrophils>0.5×109/L, platelets>25.0×109/L;
5. There is no active grade II or higher acute GVHD or moderate or severe chronic GVHD;
6. Liver and kidney function: liver function (AST/ALT/TB) <5 times normal upper limit; renal function (Cr) < 2 times normal upper limit;
7. The patient must be able to understand and be willing to participate in the study and sign an informed consent form.

Exclusion criteria:

Possible subjects who meet any of the following criteria will be excluded from the trial:

1. Recurrence after transplantation;
2. Patients who have not achieved complete remission after transplantation;
3. Implantation failed;
4. Pregnant or lactating women;
5. Have received other interventions or are receiving other research drugs before the study begins;
6. Patient blood routine: ANC <0.5 × 109 / L or PLT < 25 × 109 / L;
7. There are active uncontrolled infections: hemodynamic instability associated with infection, or new signs or signs of infection, or new infections in imaging, persistent fever with asympto or signs cannot be ruled out Infected person
8. People infected with HIV;
9. Active hepatitis B (HBV), active hepatitis C (HCV) requires antiviral therapy; patients with HBV activation risk refer to patients with hepatitis B surface antigen positive or core antibody positive patients who do not receive anti-HBV treatment;
10. Those who are allergic to known azacitidine or interferon;
11. At the discretion of the investigator, other dangerous complications may result.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2022-08-28 (Estimated); Study Completion 2022-08-28 (Estimated)

PRIMARY OUTCOMES:
Treatment response rate | 6months
  Treatment response rate after 6 months of pretreatment with azacitidine combined with interferon (primary response + secondary response)

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, M.D, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xianmin Song, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No